CLINICAL TRIAL: NCT01163305
Title: Identifying an Early Indicator of Drug Efficacy in Patients With Advanced Colorectal Cancer - a Prospective Evaluation of Circulating Tumor Cells, Positron-emission Tomography Scan and RECIST Criteria
Brief Title: PET-CT and Circulating Tumor Cells in Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CCTU, Prof. Brigette Ma, Chinese University of Hong Kong
Other Study IDs: COL016
Record Dates: First submitted 2010-06-24; First posted 2010-07-15 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Cancer; Metastasis
Keywords: Identifying an early indicator of drug efficacy
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — circulating tumor cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- metastatic colorectal cancer
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — The majority of patients offered either oxaliplatin or irinotecan-based chemotherapy

SUMMARY:
The purpose of this study is to identify an early indicator of drug efficacy in patients with advanced colorectal cancer - a prospective evaluation of circulating tumor cells, positron-emission tomography scan and RECIST criteria.

DETAILED DESCRIPTION:
1. To determine if measuring both tumor metabolic response (via FDG-PET scan) & circulating tumor cells (CirTC) at 4 weeks after starting treatment, is a better predictor of clinical outcome than measuring either modality alone in patients with metastatic colorectal cancer (CRC) who are undergoing first-line oxaliplatin-based chemotherapy.
2. To determine if a new method of assessing drug response (measuring tumor metabolic response via FDG-PET & CirTC at 4 weeks after starting treatment) better predicts clinical outcome than the conventional method (measuring radiological changes in tumor dimensions at 10 weeks after starting treatment via the 'Response Evaluation Criteria in Solid Tumors' - RECIST).

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal cancer patients not received prior drug treatment for metastatic CRC
* Age >= 18 years
* (ECOG) performance status of 0-2
* Measurable tumor sites by RECIST criteria
* Adequate bone marrow, renal & hepatic functions

Exclusion Criteria:

* Patients with diabetes mellitus
* presence of hyperglycemia
* Pregnant or lactating patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with metastatic colorectal cancer
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2010-06-30 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Tumor metabolic response via FDG-PET at 4 weeks after chemotherapy | 2 years

SECONDARY OUTCOMES:
Overall survival | 4 years
Progression-free survival | 4 years
serum carcinoembryonic antigen (CEA) level | 4 years
Circulating tumor cells level changes at 4 weeks after chemotherapy | 2 years
RECIST-based tumor response at 10 weeks after chemotherapy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Brigette Ma, MD, FRCP, Principal Investigator — Department of Clinical Oncology, Prince of Wales Hospital, The Chinese University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong